CLINICAL TRIAL: NCT04065373
Title: ivWatch SmartTouch Sensor: Device Validation for Non-Infiltrated Tissues
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ivWatch, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IVW-CLR-CS24-400
Record Dates: First submitted 2019-08-20; First posted 2019-08-22 (Actual); Last update posted 2019-08-22 (Actual); Status verified 2019-08

CONDITIONS: Infiltration of Peripheral IV Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Non-Infiltrated Tissue (Experimental): The ivWatch Model 400 with SmartTouch or fiber optic sensor monitored a common peripheral IV site over a 24 hour observation period.
  Interventions: Device: ivWatch Model 400 with SmartTouch and fiber optic sensor

INTERVENTIONS:
Device: ivWatch Model 400 with SmartTouch and fiber optic sensor — The ivWatch Model 400 with SmartTouch or fiber optic sensor monitored tissue at common IV sites over a 24 hour period.

SUMMARY:
A single arm study of 40 adult volunteers to assess the safety and efficacy of the ivWatch SmartTouch and fiber optic sensors when observing non-infiltrated (normal) tissues at common peripheral IV therapy sites.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Pass health screen
* 18 years or older

Exclusion Criteria:

* Fail health screen

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2019-04-25 (Actual); Primary Completion 2019-06-21 (Actual); Study Completion 2019-06-21 (Actual)

PRIMARY OUTCOMES:
Normal Tissue Red Notification Rate | 24 Hours
  The ivWatch Model 400 issues red notifications to communicate the need for a clinician to check an IV site. A red notification suggests an increased likelihood that an IV infiltration may be occurring, with a greater likelihood relative to a yellow notification. This measure describes the average number of red notifications issued by the ivWatch device in a given day when monitoring normal, non-infiltrated tissues. The 95% confidence interval for the red notification rate was calculated using a negative binomial regression model.

SECONDARY OUTCOMES:
Normal Tissue Yellow Notification Rate | 24 Hours
  The ivWatch Model 400 issues yellow notifications to communicate the need for a clinician to check an IV site. A yellow notification suggests an increased likelihood that an IV infiltration may be occurring, although at a lower likelihood relative to a red notification. This measure describes the average number of yellow notifications issued by the ivWatch device in a given day when monitoring normal, non-infiltrated tissues. The 95% confidence interval for the yellow notification rate was calculated using a negative binomial regression model.
Significant Skin Irritation or Disruption to Skin Integrity | 24 Hours
  The number of IV sites with significant skin irritation or disruption to skin integrity assessed at the end of the study. The Clopper-Pearson method was used for estimating the binomial proportion confidence interval.

CONTACTS AND LOCATIONS:
Overall Officials: Marisa Cole, Study Director — Employee
Locations (1):
- ivWatch, LLC, Williamsburg, Virginia, United States